CLINICAL TRIAL: NCT07356856
Title: Efficacy and Safety of Microtransplantation for Advanced and Relapsed Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Principal Investigator, xiang lu, Director, The Affiliated Hospital of the Chinese Academy of Military Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MST-ST-02
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Advanced and Relapsed Solid Tumors
Keywords: microtransplantation; solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- microtransplantation; MST (Experimental): conventional chemotherapy with microtransplantation
  Interventions: Biological: MST

INTERVENTIONS:
Biological: MST — conventional chemotherapy with microtransplantation(MST). Microtransplantation, which is the infusion of granulocyte colony stimulating factor (G-CSF) mobilized HLA-mismatched peripheral blood mononuclear cells (GPBMC)

SUMMARY:
In this study, microtransplantation (MST) will be administrated to patients diagnosed with advanced / relapsed solid tumors to assess the therapeutic efficacy and safety of conventional chemotherapy in combination with MST for the treatment of advanced/relapsed solid tumors.

DETAILED DESCRIPTION:
In this study, the eligible patients will receive MST treatment following conventional chemotherapy, MST is the infusion of G-PBMCs after chemotherapy. G-PBMCs are peripheral blood mononuclear cells from HLA mismatched unrelated donors mobilized by granulocyte colony-stimulating factor (G-CSF).

Based on the patient's medical history, current tumor assessment results, and the latest cancer treatment guidelines, an individualized chemotherapy plan for the patient is formulated through discussions among more than three oncologists. After each course of treatment, all relevant indicators, including efficacy and safety measures are evaluated.

Patients will receive all treatment for four courses, with an interval of 21 to 28 days. After completing all the treatment courses, the patient will enter the evaluation stage. Patients who have entered the evaluation stage are permitted to receive any treatments, including symptomatic support treatment, after the completion of treatment or withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients are 18 to 90 years old, regardless of gender or race;
* Advanced / relapsed solid tumors (small cell lung cancer, ovarian cancer, cervical cancer, gastric and colorectal cancer, sarcoma, head and neck tumor, etc.) are confirmed by clinical or histopathological diagnosis;
* More than two kinds of tumors are allowed;
* Karnofsky score ≥ 40, ECoG physical status ≤ 3;
* There are measurable lesions;

Exclusion Criteria:

* The researchers considered patients who were not suitable to participate in this experiment；
* Patients with mental disorders；
* Patients who refuse to cooperate with the treatment；

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-01-16 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events | 1 month
  Treatment related mortality
time of hematopoietic recovery | 1 month
  Absolute neutrophil count >500/μL; Platelets ≥20,000/μL

SECONDARY OUTCOMES:
Disease Control Rate, DCR | 1 year
  (markedly effective + effective + stable disease) / number of patients × 100%

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Lu, Professor, Principal Investigator — The First People's Hospital of Nanning; huiqin Wei, Professor, Principal Investigator — Minzu Hospital of Guangxi Zhuang Autonomous Region; yajing Huang, Professor, Principal Investigator — Innovvy(Beijing) Biomedical Technology Co., Ltd
Locations (3):
- China (3):
  - Innovvy(Beijing) Biomedical Technology Co., Ltd, Haidian, Beijing Municipality
  - Minzu Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The First People's Hospital of Nanning, Nanning, Guangxi

IPD SHARING:
Plan to Share IPD: No